CLINICAL TRIAL: NCT02012842
Title: The Effect of Periodontal Treatment on Quality of Life in Patients With Metabolic Syndrome
Brief Title: Metabolic Syndrome and Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Patricia Weidlich, Patricia Weidlich, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 060173
Record Dates: First submitted 2013-10-30; First posted 2013-12-16 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome; Periodontal Disease; Inflammatory Response
Keywords: Metabolic Syndrome; Periodontal Disease; Periodontal therapy; inflammatory markers; C reactive protein; serum fibrinogen; glycated hemoglobin
MeSH Terms: conditions — Metabolic Syndrome; Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate periodontal treatment (Active Comparator): Strict supragingival plaque control and non surgical periodontal treatment immediately after the baseline examination(test group).
  Interventions: Other: Non surgical periodontal treatment
- Delayed periodontal treatment (Other): Strict plaque control and non surgical periodontal treatment 6 months after the baseline examination (control group).
  Interventions: Other: Non surgical periodontal treatment

INTERVENTIONS:
Other: Non surgical periodontal treatment — Treatment of gingivitis: excavation and sealing of cavities, removal of overhanging restorations, extraction of hopeless teeth, supragingival calculus removal. Oral hygiene instruction, training and motivation will be given at each appointment. Treatment of periodontitis: subgingival scaling and root planing under local anesthesia.
  Other Names: strict supragingival plaque control; non surgical periodontal therapy; scaling and root planning

SUMMARY:
The aim of this study is to evaluate the effect of periodontal treatment on systemic inflammation and quality of life of individuals with metabolic syndrome. There will be a randomized clinical trial with patients from the clinic of Endocrinology - Prediabetes (Hospital de Clinicas de Porto Alegre) and outpatient dental clinic of the Faculty of Dentistry, Federal University of Rio Grande do Sul (UFRGS), who have a diagnosis of metabolic syndrome and diagnosis of periodontitis. The clinical trial will consist of an arm where it will be immediately periodontal treatment (test group) and another arm which will be held later periodontal treatment (control group). The study will last six months , and after this period, the control group will receive the same treatment to the test group . A socio-demographic questionnaire will be applied by a trained interviewer , so that data on income, education , behavioral habits , medical and dental history . Complete periodontal examination will be conducted at 6 sites per tooth for all teeth present at baseline and 3 and 6 months after periodontal treatment . In addition to the tests required for the diagnosis of metabolic syndrome , will be asked the same blood tests at 3 and 6 months after periodontal treatment (total cholesterol , LDL and HDL , fasting glucose , triglycerides , C-reactive protein). Aliquots of plasma from blood collected in each experimental point are stored at -80 ° C for analysis of interleukin- 6, Tumor Necrosis Factor- α (TNF-α) , Glucagon Like Peptide-1 (GLP-1) and adiponectin. At each clinical examination will be collected gingival crevicular fluid , supra and subgingival biofilm . Versions of the questionnaires validated in Brazil (OHIP-14)and WHOQoL Bref will be applied to assess quality of life at baseline and after 6 months of the study . The primary outcome will be change in glycated hemoglobin and secondary outcomes will be changes in serum fibrinogen and C-reactive protein.The hypothesis of this study considers that periodontal treatment can alter the serum levels of C-reactive protein, fibrinogen and glycosylated hemoglobin in patients with metabolic syndrome and thereby contribute to improved quality of life. The objective of this study is to evaluate the effect of periodontal treatment on systemic inflammation and quality of life of individuals with metabolic syndrome.

DETAILED DESCRIPTION:
There will be a randomized clinical trial with patients from the outpatient clinic of Endocrinology - Prediabetes and outpatient dental clinic of the Faculty of Dentistry, UFRGS who have a diagnosis of metabolic syndrome and diagnosis of periodontitis. The clinical trial will consist of an arm where it will be immediately periodontal treatment (test group) and another arm which will be held later periodontal treatment (control group). The study will last for six months , and after this period, the control group will receive the same treatment to the test group .

A socio-demographic questionnaire will be applied by a trained interviewer , so that data on income, education , behavioral habits , medical and dental history. A questionnaire with some key questions will be repeated in 10 % of the sample within seven days after the first application in order to check the reproducibility of the instrument.

Complete periodontal examination will be conducted at 6 sites per tooth for all teeth present at baseline and 3 and 6 months after periodontal treatment. The examination will be conducted by two examiners trained and calibrated. There will be measured Probing Depth , Bleeding On Probing, Periodontal Attachment Loss , Gingival Bleeding Index , Visible Plaque Index and the retentive factors of plaque.

In addition to the tests required for the diagnosis of metabolic syndrome , will be did the same blood tests at 3 and 6 months after periodontal treatment (total cholesterol , LDL and HDL , fasting glucose , triglycerides , C-reactive protein) . Aliquots of plasma from blood collected in each experimental point are stored at -80 ° C for analysis of interleukin- 6, TNF- α , GLP-1 and adiponectin .

At each clinical examination will be collected gingival crevicular fluid , and subgingival biofilm above 4 sites randomized among those with higher probing depth at baseline. The sites of fluid collection will be properly insulated with cotton rolls and / or gauze and dried with air jets . From the introduction of rectangles of absorbent paper (Periopaper ) for 30 seconds will be held in the gingival sulcus fluid collection . Periopaper strips are analyzed for volume (Periotron 8000) and stored in sterile plastic tube at -80 ° C until analysis. The presence of Il- 1β , IL-6 and TNF- α in the gingival fluid will be identified by flow cytometry .

The supragingival plaque will be collected with sterile spoon dentin and subgingival plaque will be collected with a sterile paper cone inserted in selected sites for 30 seconds , after drying the surface and careful removal of supragingival plaque . The cones are stored in sterile plastic tube at -80 ° C until analysis. The identification of total bacterial load and microbial periodontal ( Porphyromonas gingivalis , Fusobacterium nucleatum , Prevotella intermedia and Streptpcoccus mitis ) will be performed using the technique of real -time PCR and T - RFLP .

Dental treatment will be performed by two periodontists who either ignore the data for examination of patients . The test group will receive nonsurgical periodontal treatment in 4 weeks. The treatment will include caries removal and sealing of cavities or caries restoration , removal of restorations maladaptive , extraction of residual roots , removal of supragingival calculus and subgingival scaling and root planing under local anesthesia . Instruction, training and motivation for oral hygiene will be addressed throughout treatment. Completed treatment , patients return to fortnightly visits to the 3 month and monthly until month 6 , where it will be professional removal of supra and subgingival biofilm , and oral hygiene instruction . In 3 and 6 months will also be repeated full mouth examination for both test and control groups .

The control group will receive information about periodontal disease, as well as an oral hygiene kit consisting of multicerdas toothbrush , toothpaste and interdental brush . The same treatment given to the test group will be held in the control group immediately after the 6-month assessment . The period of six months waiting for dental treatment for individuals in the control group is supported in the literature

ELIGIBILITY:
Inclusion Criteria:

* older than or equal to 18
* at least 10 teeth
* diagnosis of periodontitis ( > 2 interproximal sites with PD> 5 mm in distinct teeth or > 2 interproximal sites with PI > 4mm in different teeth of according to Page and Eke , 2007)
* have metabolic syndrome (The patient must present at least among the following three criteria: (a ) waist circumference greater than 90 inches for men and for women over 80 , (b) triglycerides ≥ 150 mg / dl ( 1.7 mmol / L ) or as a treatment for hypertriglyceridemia (c ) HDL cholesterol less than 40 mg / dL for men and less than 50 mg / dl for women or being treated for dyslipidemia ; ( d ) hypertension at examination ( systolic ≥ 130 mm Hg and diastolic blood pressure ≥ 85 mm Hg ) or hypertension diagnosis or past history or treatment for hypertension , (e ) plasma glucose ≥ 100 mg / dl or a diagnosis of diabetes or use of medication for glycemic control)

Exclusion Criteria:

* have periodontal treatment performed in the last six months
* have used antibiotics in the last 3 months
* have indication of antibiotic prophylaxis for dental care
* be pregnant
* chronic use of systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes at glycated hemoglobin. | This measure will be measured in 0 (baseline), 3 and 6 months after periodontal treatment.
  Glycated hemoglobin will be measured by collecting blood tests at 0, 3 and 6 months after the periodontal treatment (test and control)

SECONDARY OUTCOMES:
Changes at Protein C reactive and serum fibrinogen. | These outcomes will be measured at 0, 3 and 6 months after periodontal treatment.
  Protein C reactive and serum fibrinogen will be measured by collecting blood tests at 0, 3 and 6 months after the periodontal treatment (test and control).

CONTACTS AND LOCATIONS:
Overall Officials: Rui V Oppermann, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Fernando Gerchman, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Faculty of Dentistry, Federal University of Rio Grande do Sul and Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Faculdade de Odontologia da UFRGS, Porto Alegre, Rio Grande do Sul